CLINICAL TRIAL: NCT06846268
Title: Phase II Trial of Neoadjuvant ADG126 and Pembrolizumab in Locally Advanced Colorectal Cancer
Brief Title: Neoadjuvant ADG126 and Pembrolizumab in Locally Advanced Colorectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Collaborators: Adagene Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CR01/01/24
Record Dates: First submitted 2025-02-24; First posted 2025-02-26 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Locally Advanced Colorectal Cancer
Keywords: ADG126; Pembrolizumab; Colorectal cancer; Neoadjuvant
MeSH Terms: conditions — Colorectal Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: A safety run-in phase will be performed before dose expansion at the designated dose level.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ADG126 in combination with pembrolizumab (Experimental): ADG 126 will be administered with Pembrolizumab on Day 1 and Day 22 or Pembrolizumab on Day 22 alone depending on the dose level.
  Interventions: Drug: ADG126; Drug: Pembrolizumab

INTERVENTIONS:
Drug: ADG126 — Administered via intravenous infusion on Day 1 only (Q6W) or Day 1 and Day 22 (Q3W).
Drug: Pembrolizumab — Administered via intravenous infusion on Day 1 and Day 22.
  Other Names: Keytruda

SUMMARY:
This is a single site, open-label, single-arm phase II study to determine feasibility, tolerability, and preliminary efficacy of neoadjuvant ADG126 and pembrolizumab in stage II or III colorectal cancer.

DETAILED DESCRIPTION:
This clinical trial aims to enrol patients with stage II or III colorectal cancer. At least 16, and up to 20 patients will be recruited. Patients will be given two cycles of neoadjuvant immunotherapy (ADG 126 and pembrolizumab). They will be assessed for response at 4 weeks or if they develop clinical symptoms of progression. Patients will undergo surgery 2 weeks (± 1 week) after the second dose of study treatment and within 8 weeks of study enrolment.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent for the trial.
2. Be ≥ 21 years of age on the date of signing informed consent.
3. ECOG performance status of 0 or 1.
4. Histologically confirmed colorectal adenocarcinoma. Rectal cancers allowed if the treatment plan was upfront surgery with no need for any neoadjuvant chemotherapy or radiation.
5. Clinical stage II (T3-4, N-) or stage III (Tany, N+).
6. No evidence of distant metastases.
7. Radiologically measurable or clinically evaluable disease.
8. Negative pregnancy test done 72 hours before registration, for women of childbearing potential.

   Subjects of childbearing potential must be willing to use an adequate method of contraception. Appropriate methods of birth control include abstinence, oral contraceptives, implantable hormone contraceptives, or double barrier method (diaphragm plus condom). Contraception, for the course of the study starting with the first dose of study medication through 150 days after the last dose of study medication. Note: abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

   Non-childbearing potential is defined as follows:
   * ≥45 years of age and has not had a menstrual period for >1 year
   * Patients who have been amenorrhoeic for <2 years without a history of hysterectomy and oophorectomy must have a follicle-stimulating hormone value in the postmenopausal range upon screening evaluation
   * Post-hysterectomy, post-bilateral oophorectomy, or post-tubal ligation. Documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by ultrasound. Tubal ligation must be confirmed with medical records of the actual procedure; otherwise, the patient must be willing to use 2 adequate barrier methods throughout the study.
9. Demonstrate adequate organ function as defined below, all screening labs should be performed within 28 days of treatment initiation.

   1. Haematological

      * Absolute neutrophil count (ANC) greater than or equal to 1,500/mcL.
      * Platelets greater than or equal to 100,000/mcL.
      * Haemoglobin greater than or equal to 9 g/dL.
   2. Renal

      · Serum creatinine OR Measured or calculated creatinine clearance (by Cockcroft-Gault equation), Serum creatinine less than or equal to 1.5 x upper limit of normal (ULN) OR creatinine clearance greater than or equal to 60 mL/min for subject with creatinine levels greater than 1.5 x ULN
   3. Hepatic

      * Serum total bilirubin less than or equal to 1.5 x ULN OR Direct bilirubin less than or equal to ULN for subjects with total bilirubin levels greater than 1.5 x ULN.
      * AST and ALT less than or equal to 2.5 x ULN.
   4. Coagulation · International Normalised Ratio (INR) or Prothrombin Time (PT) or Activated Partial Thromboplastin Time (aPTT). For patients not taking warfarin: INR less than or equal to 1.5 or PT less than or equal to 1.5 x ULN; and either PTT or aPTT less than or equal to 1.5 x ULN. Patients on warfarin may be included on a stable dose with a therapeutic INR less than 3.5.

Exclusion Criteria:

1. Recurrent colorectal cancer.
2. Prior radiation therapy, chemotherapy, immunotherapy, or surgery for colorectal cancer.
3. Tumour is causing symptomatic bowel obstruction (patients who have a temporary diverting stoma are eligible).
4. Other invasive malignancy ≤5 years prior to registration.
5. Diagnosis of immunodeficiency or receiving systemic steroid therapy or any other form of non-physiologic dose immunosuppressive therapy within 7 days prior to first dose of trial treatment.
6. Active autoimmune disease requiring systemic treatment within the past 2 years or documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents at non-physiologic doses.
7. Active infection requiring systemic therapy.
8. Received prior therapy with an antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways.
9. Experienced ≥ Grade 3 immune-related adverse event with prior immunotherapy, with the exception of non-clinically significant lab abnormalities.
10. Other anticancer or experimental therapy. No other experimental therapies (including chemotherapy, radiation, hormonal treatment, antibody therapy, immunotherapy, gene therapy, vaccine therapy, angiogenesis inhibitors, or other experimental drugs) of any kind are permitted while the patient is receiving study treatment.
11. Known history of Human Immunodeficiency Virus.
12. Known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
13. Women who are pregnant or breastfeeding, or men expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening visit through 150 days after the last dose of study medication.
14. Concurrent medical or psychiatric condition or disease which, in the investigator's judgement, would make them inappropriate candidates for entry into the study. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 90 days) myocardial infarction, chronic obstructive pulmonary disease, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, or any psychiatric disorder that prohibits obtaining informed consent.
15. Received a live vaccine within 30 days of planned start of study medication.
16. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to enrolment.
17. History of interstitial lung disease.
18. Known hypersensitivity to ADG126 or pembrolizumab components or excipients.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04-14 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of Major Pathologic Response (MPR) | Up to 4 months
  MPR is defined as less than or equal to 10% of residual viable tumour in the surgical specimen.

SECONDARY OUTCOMES:
Rate of Pathologic Complete Response (pCR) | Up to 4 months.
  pCR is defined as the absence of any residual viable tumour in the surgical specimen.
Objective Response Rate (ORR) | Up to 4 months.
  Determined by the investigator according to RECIST 1.1 criteria.
Disease-free survival (DFS) | Up to 5 years from surgery.
  DFS is defined as the time from surgery to the first occurrence of disease relapse or death from any cause.
Adverse Events and Serious Adverse Events | From screening to 30 days after last day of study participation.
  Graded using NCI CTCAE toxicity grading v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Wei Peng Yong, MD, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Background] Alieva M, van Rheenen J, Broekman MLD. Potential impact of invasive surgical procedures on primary tumor growth and metastasis. Clin Exp Metastasis. 2018 Apr;35(4):319-331. doi: 10.1007/s10585-018-9896-8. Epub 2018 May 4. PMID 29728948
- [Background] Andre T, Shiu KK, Kim TW, Jensen BV, Jensen LH, Punt C, Smith D, Garcia-Carbonero R, Benavides M, Gibbs P, de la Fouchardiere C, Rivera F, Elez E, Bendell J, Le DT, Yoshino T, Van Cutsem E, Yang P, Farooqui MZH, Marinello P, Diaz LA Jr; KEYNOTE-177 Investigators. Pembrolizumab in Microsatellite-Instability-High Advanced Colorectal Cancer. N Engl J Med. 2020 Dec 3;383(23):2207-2218. doi: 10.1056/NEJMoa2017699. PMID 33264544
- [Background] Argiles G, Tabernero J, Labianca R, Hochhauser D, Salazar R, Iveson T, Laurent-Puig P, Quirke P, Yoshino T, Taieb J, Martinelli E, Arnold D; ESMO Guidelines Committee. Electronic address: clinicalguidelines@esmo.org. Localised colon cancer: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2020 Oct;31(10):1291-1305. doi: 10.1016/j.annonc.2020.06.022. Epub 2020 Jul 20. No abstract available. PMID 32702383
- [Background] Blank CU, Lucas MW, Scolyer RA, van de Wiel BA, Menzies AM, Lopez-Yurda M, Hoeijmakers LL, Saw RPM, Lijnsvelt JM, Maher NG, Pulleman SM, Gonzalez M, Torres Acosta A, van Houdt WJ, Lo SN, Kuijpers AMJ, Spillane A, Klop WMC, Pennington TE, Zuur CL, Shannon KF, Seinstra BA, Rawson RV, Haanen JBAG, Ch'ng S, Naipal KAT, Stretch J, van Thienen JV, Rtshiladze MA, Wilgenhof S, Kapoor R, Meerveld-Eggink A, Grijpink-Ongering LG, van Akkooi ACJ, Reijers ILM, Gyorki DE, Grunhagen DJ, Speetjens FM, Vliek SB, Placzke J, Spain L, Stassen RC, Amini-Adle M, Lebbe C, Faries MB, Robert C, Ascierto PA, van Rijn R, van den Berkmortel FWPJ, Piersma D, van der Westhuizen A, Vreugdenhil G, Aarts MJB, Stevense-den Boer MAM, Atkinson V, Khattak M, Andrews MC, van den Eertwegh AJM, Boers-Sonderen MJ, Hospers GAP, Carlino MS, de Groot JB, Kapiteijn E, Suijkerbuijk KPM, Rutkowski P, Sandhu S, van der Veldt AAM, Long GV. Neoadjuvant Nivolumab and Ipilimumab in Resectable Stage III Melanoma. N Engl J Med. 2024 Nov 7;391(18):1696-1708. doi: 10.1056/NEJMoa2402604. Epub 2024 Jun 2. PMID 38828984
- [Background] Cercek A, Lumish M, Sinopoli J, Weiss J, Shia J, Lamendola-Essel M, El Dika IH, Segal N, Shcherba M, Sugarman R, Stadler Z, Yaeger R, Smith JJ, Rousseau B, Argiles G, Patel M, Desai A, Saltz LB, Widmar M, Iyer K, Zhang J, Gianino N, Crane C, Romesser PB, Pappou EP, Paty P, Garcia-Aguilar J, Gonen M, Gollub M, Weiser MR, Schalper KA, Diaz LA Jr. PD-1 Blockade in Mismatch Repair-Deficient, Locally Advanced Rectal Cancer. N Engl J Med. 2022 Jun 23;386(25):2363-2376. doi: 10.1056/NEJMoa2201445. Epub 2022 Jun 5. PMID 35660797
- [Background] Morton D, Seymour M, Magill L, Handley K, Glasbey J, Glimelius B, Palmer A, Seligmann J, Laurberg S, Murakami K, West N, Quirke P, Gray R; FOxTROT Collaborative Group. Preoperative Chemotherapy for Operable Colon Cancer: Mature Results of an International Randomized Controlled Trial. J Clin Oncol. 2023 Mar 10;41(8):1541-1552. doi: 10.1200/JCO.22.00046. Epub 2023 Jan 19. PMID 36657089